CLINICAL TRIAL: NCT02279407
Title: A Double-blind Randomized Placebo-controlled, Parallel-group 12 Week Study to Investigate the Effects of Omega-3 Carboxylic Acids and Dapagliflozin on Liver Fat Content in Type 2 Diabetic Patients; EFFECT II
Brief Title: A Study to Investigate Effects of Omega-3 Carboxylic Acids and Dapagliflozin on Liver Fat Content in Diabetic Patients
Acronym: EFFECTII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Uppsala Clinical Research, Uppsala, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5883C00004
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: T2 Diabetes and Fatty Liver Disease (Non-alcoholic Origin)
Keywords: omega-3 carboxylic acid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Omega-3 carboxylic acids 4g / day (Experimental)
  Interventions: Drug: Omega-3 carboxylic acids
- Dapagliflozin, 10mg / day (Experimental)
  Interventions: Drug: Dapagliflozin
- Omega-3 carboxylic acids 4g/day+Dapagliflozin 10mg/day (Experimental)
  Interventions: Drug: Omega-3 carboxylic acids; Drug: Dapagliflozin

INTERVENTIONS:
Drug: placebo — Placebo matching to Omega-3 carboxylic acids (olive oil)
  Arms: placebo
Drug: Omega-3 carboxylic acids — 4 g administered as 4 x 1 g capsules
  Arms: Omega-3 carboxylic acids 4g / day; Omega-3 carboxylic acids 4g/day+Dapagliflozin 10mg/day
Drug: Dapagliflozin — 10 mg administered as 10 mg tablet
  Arms: Dapagliflozin, 10mg / day; Omega-3 carboxylic acids 4g/day+Dapagliflozin 10mg/day
Drug: Placebo — Placebo matching to dapagliflozin 10 mg
  Arms: placebo

SUMMARY:
This study is a double-blind randomized, placebo-controlled, parallel-group, 12 week study performed in up to 5 centres in Sweden to assess the effect of Omega-3 carboxylic acids and dapagliflozin on liver fat in patients with Type 2 diabetes with fatty liver (>5.5% as measured with magnetic resonance imaging (MRI))

ELIGIBILITY:
Inclusion Criteria: Provision of informed consent prior to any study specific procedures; Men or women ≥40 years and ≤75 years with suitable veins for cannulation or repeated venepuncture; Have liver fat content as assessed by MRI >5.5%; Diagnosis of Type 2 diabetes since at least 6 months in accordance with WHO criteria.

Exclusion Criteria: Any condition when MRI is contraindicated such as, but not limited to, having a pacemaker or claustrophobia; Diagnosis or signs of Type 1 diabetes (e.g. history of positive islet antibodies); Creatinine clearance <60 mL/min at screening (Cockcroft-Gault formula).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eriksson, MD, Principal Investigator — Uppsala University Hospital, Uppsala, SE
Locations (5):
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Eriksson JW, Lundkvist P, Jansson PA, Johansson L, Kvarnstrom M, Moris L, Miliotis T, Forsberg GB, Riserus U, Lind L, Oscarsson J. Effects of dapagliflozin and n-3 carboxylic acids on non-alcoholic fatty liver disease in people with type 2 diabetes: a double-blind randomised placebo-controlled study. Diabetologia. 2018 Sep;61(9):1923-1934. doi: 10.1007/s00125-018-4675-2. Epub 2018 Jul 3. PMID 29971527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 centers in Sweden between 20 January 2015 and 11 December 2015.
Pre-assignment Details: The study duration was up to 15 weeks: an screening period of up to 2 weeks, a 12-week treatment period, and a follow-up visit 1 week after the last dose of study drug. A total of 223 patients signed informed consent; data was not recorded for 1 patient and 18 were screened twice. Therefore, 204 patients were screened, and 84 were randomized.
Groups:
- Epanova + Dapagliflozin: Epanova 4 g/day + Dapagliflozin 10 mg/day
- Dapagliflozin: Dapagliflozin 10 mg/day + placebo to Epanova
- Epanova: Epanova 4 g/day + placebo to Dapagliflozin
- Placebo: Placebo to Epanova and placebo to Dapagliflozin
Period: Overall Study
Arm/Group | Epanova + Dapagliflozin | Dapagliflozin | Epanova | Placebo
Started | 22 | 21 | 20 | 21
Completed | 20 | 20 | 15 | 20
Not Completed | 2 | 1 | 5 | 1
Not completed — Couldn't swallow IP; noncompliance | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epanova + Dapagliflozin | Epanova | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 21 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (5.42) [54 to 74] | 66.2 (5.94) [50 to 73] | 65.0 (6.54) [48 to 74] | 65.6 (6.10) [52 to 74] | 65.5 (5.92) [48 to 74]
Age, Customized [Number; unit: Participants]
  <50 | 0 | 0 | 1 | 0 | 1
  >=50 - <65 | 9 | 6 | 6 | 6 | 27
  >=65 | 13 | 14 | 14 | 15 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 5 | 4 | 25
  Male | 15 | 11 | 16 | 17 | 59
Race/Ethnicity, Customized [Number; unit: Participants]
  Black Or African American | 1 | 0 | 1 | 0 | 2
  White | 21 | 20 | 20 | 21 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in % Liver Fat as Assessed by MRI (Comparison Versus Placebo)
Description: To evaluate the efficacy of the combination therapy (Epanova + Dapagliflozin) when compared to placebo with respect to reduction in liver fat content (%) at the end of 12 weeks of double-blinded treatment. Treatment effect in liver fat reduction (%) was assessed using a mixed linear model with the change from baseline on logarithmic scale as response variable and the logarithm of the baseline value as covariate, treatment as fixed effect, and center as random effect. The treatment effect was then back-transformed to original scale as Geometric mean ratio and presented as percentage change from baseline.
Time Frame: 12 weeks
Population: The Full Analysis Set included all randomized patients, regardless of whether they took trial medication or not. In this set, patients were analyzed according to their randomized treatment assignment.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of % liver fat
Arm/Group | Epanova + Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 19
ratio of % liver fat | 0.79 [0.69 to 0.90] | 0.97 [0.90 to 1.04]
Statistical Analysis 1: Comparison: Epanova + Dapagliflozin vs Placebo; Test type: Superiority or Other; p = 0.046, Mixed Models Analysis — Hypotheses tested using Dunnett's multiple testing procedure with a family-wise error rate of 5%, adjusting for 3 pairwise comparisons versus a single control (placebo); Geometric mean ratio for difference = 0.83, 95% CI 2-sided [0.70 to 1.00]

2. Secondary Outcome: Change From Baseline to Week 12 in % Liver Fat (Comparison Between Active Treatment Groups)
Description: To evaluate the relative efficacy of the combination of Epanova and dapagliflozin versus Epanova alone and dapagliflozin alone with respect to reduction in % liver fat at the end of 12 weeks of double-blind treatment. Treatment effect in liver fat reduction (%) was assessed using a mixed linear model with the change from baseline on logarithmic scale as response variable and the logarithm of the baseline value as covariate, treatment as fixed effect, and center as random effect. The treatment effect was then back-transformed to original scale as Geometric mean ratio and presented as percentage change from baseline.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of % liver fat
Arm/Group | Epanova + Dapagliflozin | Dapagliflozin | Epanova
Number analyzed (Participants) | 20 | 19 | 15
ratio of % liver fat | 0.79 [0.69 to 0.90] | 0.87 [0.77 to 0.99] | 0.85 [0.78 to 0.92]
Statistical Analysis 1: Comparison: Epanova + Dapagliflozin vs Dapagliflozin; Test type: Superiority or Other; p = 0.502, Mixed Models Analysis — Conditional upon rejection of at least 1 of the 3 hypotheses for the primary analysis, secondary hypotheses are tested using Tukey's multiple testing procedure with a family-wise error rate of 5%, adjusting for 3 pairwise comparisons; Geometric mean ratio for difference = 0.91, 95% CI 2-sided [0.75 to 1.11]
Statistical Analysis 2: Comparison: Epanova + Dapagliflozin vs Epanova; Test type: Superiority or Other; p = 0.562, Mixed Models Analysis — Conditional upon rejection of at least 1 of the hypotheses for the primary analysis, secondary hypotheses are tested using Tukey's multiple testing procedure with a family-wise error rate of 5%, adjusting for 3 pairwise comparisons; Geometric mean ratio for difference = 0.91, 95% CI 2-sided [0.73 to 1.13]

ADVERSE EVENTS:
Arm/Group | Epanova + Dapagliflozin | Epanova | Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 14/22 | 12/20 | 8/21 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova + Dapagliflozin (N=22) | Epanova (N=20) | Dapagliflozin (N=21) | Placebo (N=21)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova + Dapagliflozin (N=22) | Epanova (N=20) | Dapagliflozin (N=21) | Placebo (N=21)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 7 (7) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No